CLINICAL TRIAL: NCT02416882
Title: Exercise Genes: Genomic Association With Exercise Reinforcement
Acronym: ExGenes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GFHNRC405
Record Dates: First submitted 2015-04-02; First posted 2015-04-15 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Overweight; Obesity; Physical Activity
Keywords: active; not active; normal body weight
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Exercise vs Sedentary Option (Other): Relative Reinforcing Value of aerobic exercise versus sedentary activity will be determined.
  Interventions: Other: Aerobic Exercise; Other: Sedentary Option
- Resistance Exercise vs Sedentary Option (Other): Relative Reinforcing Value of resistance exercise versus sedentary activity will be determined.
  Interventions: Other: Resistance Exercise; Other: Sedentary Option

INTERVENTIONS:
Other: Aerobic Exercise — Subjects will sample and rate their liking of three cardiovascular machines (treadmill, cycle ergometer, elliptical step ergometer) to determine which one will be used during the test.
  Arms: Aerobic Exercise vs Sedentary Option
Other: Resistance Exercise — Subjects will sample and rate their liking of three different resistance training circuits (upper body, lower body, core) to determine which one will be used during the test.
  Arms: Resistance Exercise vs Sedentary Option
Other: Sedentary Option — Subjects will rate their liking of three sedentary activities (reading magazines, playing puzzles, completing word games) as an alternative to exercise.

SUMMARY:
This study tests whether different physical activity patterns are linked an individual's genes.

DETAILED DESCRIPTION:
The investigators propose that an individual's genetics are one factor that may be associated with the motivating aspect or attractiveness of exercise and therefore the choice to exercise rather than be sedentary. They propose to study the association of the genomic signatures with the reinforcing (motivating) value of different types of exercise. This has never been investigated and may uncover underlying mechanisms that would help to understand individual differences in exercise motivation. The ultimate impact of this work is a greater number of Americans being physically active, meeting the United States Department of Agriculture (USDA) dietary guidelines for physical activity, and maintaining a healthy body weight. This study will be funded and undertaken at the Grand Forks Human Nutrition Research Center (GFHNRC). The purpose will be to assess genetic underpinnings of the motivating value of resistance and aerobic exercise, and to determine whether the motivating value of aerobic and resistance exercise are associated with usual participation in these modes of exercise.

ELIGIBILITY:
Inclusion Criteria:

* BMI within 18.5-35.0 kg/m2
* Healthy enough to exercise
* Active or inactive (not exercising at this time)

Exclusion Criteria:

* Taking any drugs that affect energy expenditure (e.g., thyroid, glucose-lowering drugs)
* Have gained or lost more than 5% of body weight over the past 6 months
* Use tobacco
* Pregnant or lactating or plan to become pregnant in the next 6 months
* Have any health conditions that prevent the individual from safely exercising (e.g., cardiovascular, liver, endocrine, or pulmonary diseases)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Relative reinforcing value (RRV) of physical activity | Week 0 (Cross-sectional)
  RRV of physical activity will be assessed by evaluating the number of responses (mouse button presses) a subject is willing to complete to gain access to physical activity or a sedentary alternative.
Preference for intense physical activity and tolerance for exercise discomfort | Week 0 (Cross-sectional)
  Preference for intense physical activity and tolerance for exercise discomfort will be assessed by self-report questionnaire responses.
Genotypes of 23 small nucleotide polymorphisms (SNPs) previously identified to influence central dopamine release or uptake, reward, or physical activity | Week 0 (Cross-sectional)
  SNP genotyping will be performed on 3-5 ml samples of whole blood collected in ethylenediaminetetraacetic acid (EDTA)-containing tubes followed by allelic-discrimination analysis for the amplification and identification of each SNP.

CONTACTS AND LOCATIONS:
Overall Officials: James N Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No